CLINICAL TRIAL: NCT07197216
Title: Evaluation of the Tap Trust Intervention on Water Security Experiences and Beverage Intake
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anisha I Patel, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 74926
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Beverage Intake; Child Health and Nutrition
Keywords: Drinking water quality; Child beverage intake; Preschoolers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants will test their home tap water using kits mailed to their homes, with phone or Zoom assistance from the research team. Families with water quality concerns will receive remediation tailored to the issue (e.g., flushing guidance, filtration device and installation guidance). Participants will also receive reusable water bottles, educational handouts and videos, and phone or Zoom sessions with the research team that include motivational interviewing to set healthy beverage goals.
  Interventions: Behavioral: Tap Trust
- Control Group (No Intervention): Participants will not receive water testing kits, filtration devices, or educational resources during the study. After the study concludes, participants will have access to the intervention materials.

INTERVENTIONS:
Behavioral: Tap Trust — Home-based intervention includes tap water testing kits (instructions provided with videos or phone/Zoom), filtration devices if water quality concerns are identified, reusable water bottles and educational materials (handouts and videos), and phone/Zoom sessions with the research team using motivational interviewing.
  Arms: Intervention Group

SUMMARY:
The primary aim of this clinical trial is to determine whether the Tap Trust intervention increases water intake among preschool-aged children and their parents/caregivers by improving families' experiences with their home tap water.

ELIGIBILITY:
Inclusion Criteria:

1. Parents/caregivers of pre-school aged children from the Healthy Drinks, Healthy Futures study childcare centers that did not receive the program.
2. Parents/caregivers must speak English or Spanish.
3. Parents/caregivers of preschool-age children who don't have health conditions that preclude intake of water.

Exclusion Criteria:

Parents/caregivers who do not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in child total plain water intake (oz/day) | Baseline and 6 months post-intervention
  Child total plain water intake assessed via validated beverage frequency questionnaires

SECONDARY OUTCOMES:
Change in child unfiltered tap water intake (oz/day) | Baseline and 6 months post-intervention
  Child unfiltered tap water intake via validated beverage frequency questionnaires
Change in child filtered tap water intake (oz/day) | Baseline and 6 months post-intervention
  Child filtered tap water intake via validated beverage frequency questionnaires
Change in child bottled water intake (oz/day) | Baseline and 6 months post-intervention
  Child bottled water intake via validated beverage frequency questionnaires
Change in child sugar-sweetened beverages (SSB) intake (oz/day) | Baseline and 6 months post-intervention
  Child SSB intake via validated beverage frequency questionnaires
Change in parent/caregiver total plain water intake (oz/day) | Baseline and 6 months post-intervention
  Parent/caregiver total plain water intake assessed via validated beverage frequency questionnaires
Change in parent/caregiver unfiltered tap water intake (oz/day) | Baseline and 6 months post-intervention
  Parent/caregiver unfiltered tap water intake via validated beverage frequency questionnaires
Change in parent/caregiver filtered water intake (oz/day) | Baseline and 6 months post-intervention
  Parent/caregiver filtered water intake via validated beverage frequency questionnaires
Change in parent/caregiver bottled water intake (oz/day) | Baseline and 6 months post-intervention
  Parent/caregiver bottled water intake via validated beverage frequency questionnaires
Change in parent/caregiver SSB intake (oz/day) | Baseline and 6 months post-intervention
  Parent/caregiver SSB intake via validated beverage frequency questionnaires
Change in parent/caregiver experience of home water security | Baseline and 6 months post-intervention
  Parent/caregiver-reported experiences using home tap water, including ratings of taste, odor, appearance, and smell from questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Anisha I Patel, MD, MSPH, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
This will need to be discussed with the community advisory board.